CLINICAL TRIAL: NCT02905110
Title: Combination Intraventricular Chemotherapy Pilot Study: Methotrexate and Etoposide Infusions Into the Fourth Ventricle or Resection Cavity in Children with Recurrent Posterior Fossa Brain Tumors
Brief Title: Methotrexate and Etoposide Infusions Into the Fourth Ventricle in Children with Recurrent Posterior Fossa Brain Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, David Ilan Sandberg, Director of Pediatric Neurosurgery, Associate Professor Pediatric Surgery and Neurosurgery, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0639
Record Dates: First submitted 2016-09-07; First posted 2016-09-19 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Brain Tumor Recurrent
Keywords: Malignant Neoplasms, Brain; medulloblastoma; ependymoma; Atypical Teratoid Rhabdoid Tumor (ATRT)
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma; Ependymoma; Rhabdoid Tumor | interventions — Methotrexate; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Methotrexate / Etoposide Infusion (Experimental): 12 infusions of intraventricular Methotrexate and 15 infusions of intraventricular Etoposide into implanted fourth ventricle catheter/Ommaya reservoir following surgical catheter placement into fourth ventricle. Methotrexate will be infused twice weekly for 6 weeks and etoposide will be infused 5 times a week on weeks 1, 3 , and 5.
  Interventions: Drug: Methotrexate; Drug: Etoposide; Procedure: Ommaya Reservoir

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 4 mg into fourth ventricle of the brain via the Ommaya Reservoir 2 days a week for 6 weeks. Each patient will have 12 infusions.
  Other Names: Trexall, Rasuvo
Drug: Etoposide — Etoposide 1 mg into fourth ventricle of the brain via the Ommaya Reservoir 5 days a week for weeks 1, 3, and 5. Each patient will have 15 infusions.
  Other Names: VePesid, Toposar, Etopophos
Procedure: Ommaya Reservoir — Surgical catheter placement into the fourth ventricle of the brain

SUMMARY:
The goal of this clinical research study is to establish the safety of simultaneous infusions of methotrexate and etoposide into the fourth ventricle of the brain or resection cavity in patients with recurrent malignant posterior fossa brain tumors. These tumors include medulloblastoma, ependymoma, atypical teratoid/rhabdoid tumor or other malignant brain tumor with recurrence or progression involving anywhere in the brain and/or spine. Patients' disease must have originated in the posterior fossa of the brain.

DETAILED DESCRIPTION:
If the participant is eligible to take part in this study, the participant will have surgery to place a catheter into the Ommaya reservoir. The Ommaya reservoir is a catheter system that allows drugs to be administered directly to parts of the brain. This catheter will be used for the infusion of methotrexate and etoposide directly into the 4th ventricle of the brain, which is 1 of the 4 connected fluid-filled cavities in the brain.

If the study doctor thinks it is necessary, based on the location of the tumor, the tumor may also be removed while the participant is already under anesthesia just before the catheter is placed.

Study Drug Administration:

The participant will receive twice weekly 4 mg intraventricular methotrexate infusions for six consecutive weeks and daily 1 mg intraventricular etoposide infusion five times per week, every 2 weeks. Etoposide will be administered on weeks 1, 3, and 5.

Methotrexate and Etoposide will be infused though the ommaya reservoir catheter directly into the 4th ventricle of the brain starting at a minimum of 7 days after the catheter placement surgery. A MRI will be done to confirm adequate cerebrospinal fluid flow. The etoposide infusion will last 3-4 minutes and the methotrexate infusion will last 3 minutes.

If the participant already has an Ommaya catheter, methotrexate and etoposide will begin after an MRI has confirmed adequate cerebrospinal fluid flow.

Study Visits:

Prior to first infusion:

Medical history will be reviewed and any updates to health will be recorded. Physical and Neurological exam with vital signs will be done. Blood (about 1 teaspoon) will be drawn for routine test. A lumbar puncture will be done. A MRI scan of the brain and spine will be done to check the status of the disease.

On the days of the Methotrexate and Etoposide Infusion:

A neurological exam with vital signs will be done. A Ommaya reservoir tap (a catheter is placed into the Ommaya reservoir to give the methotrexate and etoposide infusion.

Cerebrospinal fluid (about 1 teaspoon) will be collected for routine tests.

Within 7 days of completing the Final infusion:

A neurological exam with vital signs will be done. A lumbar puncture and lab work will be done. A MRI scan of the brain and spine will be done to check status of the disease.

Length of Study:

The participant will receive 12 infusions of Methotrexate 4 mg and 15 infusions of Etoposide 1 mg, as long as the doctor thinks it is in their best interest. The participant will no longer be able to receive the study drug if the disease gets worse, if intolerable side effects occur, or if unable to follow study directions.

This is an investigation study. Methotrexate is FDA approved and commercially available for infusion directly into brain tumors. The infusion of methotrexate into the 4th ventricle of the brain in investigational. Etoposide is FDA approved and commercially available to be given by mouth or into the bloodstream (intravenously) but has never been given in the 4th ventricle of the brain. The infusion of methotrexate and etoposide into the 4th ventricle of the brain is investigational.

Up to 10 patients will be enrolled in this study. All will be enrolled at Children's Memorial Hermann Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 - 80 years at time of recurrence or progression
* Diagnosis: Patients with histologically verified medulloblastoma, ependymoma, or atypical teratoid/rhabdoid tumor or other malignant brain tumor with recurrence or progression involving anywhere in the brain and/or spine. To be eligible, patients' disease must have originated in the posterior fossa of the brain
* Patient must have either measurable or evaluable tumor as assessed by MRI of the brain and total spine
* An implanted catheter in the fourth ventricle or posterior fossa tumor cavity attached to an Ommaya reservoir or agreement to have one placed.
* A minimum of 7 days between last dose of systemic chemotherapy and/or radiation therapy and first infusion of chemotherapy into fourth ventricle
* Life expectancy of at least 12 weeks in the opinion of the PI
* Lansky score of 50 or greater if ≤16 years of age or Karnofsky score of 50 or greater if > 16 years of age
* Existing neurological deficits must have been stable for a minimum of 1 week prior to study enrollment
* Patients must have recovered from the acute toxic effects of all prior anticancer chemotherapy
* Adequate bone marrow function defined by peripheral absolute neutrophil count (ANC) ≥ 500/µL, platelet count ≥ 50,000/µL (transfusion independent), and hemoglobin ≥ 9.0 gm/dL (may receive Red Blood Cell transfusions)
* Patient or patient's legal representative, parent(s), or guardian able to provide written informed consent.

Exclusion Criteria:

* Enrolled in another treatment protocol
* Has received another investigational or chemotherapy agent or radiation therapy within 7 days prior to intraventricular chemotherapy infusions
* Evidence of untreated infection
* Pregnant or lactating women

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with grade 3 through grade 5 new neurological adverse events that are related to study drug, graded according to NCI CTCAE Version 4.0 | 4 months
  New neurological deficit defined as new cranial neuropathy, nystagmus, change in mental status, motor deficit or cerebellar finding (ataxia, dysmetria, dysdiadochokinesis) that is attributed by treating physicians to intraventricular methotrexate and etoposide infusions. Primary endpoint for basis of safety monitoring is acute toxicity occurring at any time within 30 days of receiving the intraventricular methotrexate and etoposide infusion. Rate of acute toxicity monitored using Bayesian method of Thall and Sung. Method of Kaplan and Meier used to estimate unadjusted distributions of time to a neurological deficit and progression free survival time and summary statistic of all variable computed and tabulated

CONTACTS AND LOCATIONS:
Overall Officials: David Sandberg, MD, Principal Investigator — UTHealth
Locations (1):
- UTHealth & Children's Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No